CLINICAL TRIAL: NCT06668675
Title: Digital Intervention for School-going Adolescents: A Serious Games Approach for Cardiovascular Health Promotion in Nepal
Brief Title: Digital Cardiovascular Health Promotion Among School-going Adolescents in Nepal
Acronym: HRIDAYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu Medical College and Teaching Hospital (Other)
Collaborators: University of Skövde (Other)
Responsible Party: Principal Investigator, Dayana Shakya, Assistant Professor, Kathmandu Medical College and Teaching Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 660/2021
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Heart Disease
Keywords: Digital cardiovascular health promotion; Nepal; School-going adolescents; Mobile games; Serious games
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital intervention arm (Experimental): This intervention arm will receive the serious game known as 'Happy Heart'. The game will be installed in their mobile devices through a link. The adolescents in this arm will play the game on their mobiles for 2 weeks.
  Interventions: Other: A serious game known as the 'Happy Heart' will be used as the intervention.
- No digital intervention arm (Other): The control group adolescents will receive the same serious game 'Happy Heart' but after the study period is over
  Interventions: Other: A serious game known as the 'Happy Heart' will be used as the intervention.

INTERVENTIONS:
Other: A serious game known as the 'Happy Heart' will be used as the intervention. — The serious game known as 'Happy Heart' is a mobile game used for educational purpose in addition to entertainment. It focuses on healthy habits for the heart and is aimed at improving knowledge on diet and physical activity among school-going adolescents.
  The game is developed in collaboration with the game development team from the School of Informatics, University of Skövde and the health team from Kathmandu Medical College, Nepal.

SUMMARY:
The goal of this HRIDAYA project is to see if a digital mobile game can improve knowledge about heart disease among school-going adolescents. The researchers will divide adolescents of public and private schools into two groups. Each group will contain adolescents from both the school types. Knowledge, attitude and practice (KAP) of adolescents will be tested before intervention. One group will receive a mobile game and the other will not receive the game.

After two weeks of game play, the KAP of the adolescents will be tested again. The changes in KAP before and after playing the game in the two groups will be compared.

The participants will need to:

* Give pretest of KAP regarding CVD
* Download the game in their mobile devices.
* Install the game
* Play the game for 2 weeks
* Give post test of KAP regarding CVD

DETAILED DESCRIPTION:
With the rise in non-communicable diseases (NCDs), cardiovascular disease (CVD) prevalence is increasing in Nepal. CVD risk factors (smoking, harmful use of alcohol, insufficient intake of fruits and vegetables, obesity, hypertension, diabetes and dyslipidemia) are common among adolescents. Despite high prevalence, the knowledge, attitude and practice regarding CVD among adolescents is poor. Since CVDs often begin with modifiable risk behaviors established during adolescence which manifest later, it becomes utmost important to target this population. To tackle this growing problem, a possible way to educate the children on heart-health at the community level is through schools.

The overall aim of this HRIDAYA project is to develop a cardiovascular health education and pilot it among school-going adolescents in Nepal to improve their cardiovascular health awareness.

This HRIDAYA project is a school based parallel trial with digital health promotion intervention aimed at adolescents of grades 8-10 in the public and private schools of Jhaukhel and Duwakot Health Demographic Surveillance Site (JD-HDSS). The JD-HDSS consists of two wards Jhaukhel and Duwakot of Bhaktapur district, 13 kms away from Kathmandu, the capital of Nepal.

A baseline study was carried out to identify knowledge gaps regarding cardiovascular disease (CVDs) among adolescents. These gaps defined the learning goals of the game. Then a paper game prototype was developed in collaboration with the School of Informatics, University of Skövde, Sweden and tested among 10 adolescents. The knowledge gaps combined with the visual recognition and preferences from the paper game prototype testing were mapped into the serious game mechanics resulting in a digital serious game called 'Happy Heart'.

For the intervention, adolescents studying in grades 8-10 from one public and two private schools will be selected purposively for each of the intervention and control arm of the study. Pre-intervention testing of the knowledge, attitude and practice (KAP) will be done before the intervention. The adolescents in the intervention arm will receive a link to download the game in their mobile devices. They will play the game for 2 weeks. A post intervention test will again be done regarding the KAP for CVDs.

The data will be entered and analyzed in SPSS version 28. The change in knowledge (primary outcome), attitude and practice (secondary outcome) in the intervention and control group will be identified using the difference in difference analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents studying in grades 8-10 in public and private schools in JD-HDSS.

Exclusion Criteria:

* Adolescents absent during data collection period

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 345 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Knowledge score | 2 months
  The knowledge of the adolescents will be measured using the knowledge part of the 'Knowledge, attitude and practice of cardiovascular disease among school-going adolescents' questionnaire before and after the serious game is administered. The total knowledge score obtained by the adolescents will be converted into percentage. So the minimum score is 0% and maximum score is 100%. Higher the percent score, better will be the knowledge.
  The primary outcome is the change in knowledge score of adolescents before and after playing the serious game 'Happy Heart'.

SECONDARY OUTCOMES:
Attitude score | 2 months
  The attitude of the adolescents will be measured using the 5 point Likert scale in the attitude part of the 'Knowledge, attitude and practice of cardiovascular disease among school-going adolescents' questionnaire before and after the serious game is administered. The total score obtained by the adolescents in attitude will be converted into percentage. So the minimum score is 0% and maximum score is 100%. Higher the percent score, better will be the attitude.
  So, the secondary outcome is the change in attitude score of adolescents before and after playing the serious game 'Happy Heart'.

OTHER OUTCOMES:
Practice score | 2 months
  The practice of the adolescents will be measured using the practice part of the 'Knowledge, attitude and practice of cardiovascular disease among school-going adolescents' questionnaire before and after the serious game is administered. The practice will be scored based on the American Heart Association guidelines. These included if the adolescents ate five servings of fruits and vegetables, practiced 60 minutes of physical activity daily and did not smoke or drink.
  The total score obtained by the adolescents in practice will be converted into percentage. So the minimum score is 0% and maximum score is 100%. Higher the score better will be the practice.
  Another secondary outcome is the change in practice score of adolescents before and after playing the serious game 'Happy Heart'.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Krettek, PhD, Study Chair — University of Skövde
Locations (1):
- Kathmandu Medical College, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available after the trial results have been published.
Time Frame: IPD will be available after the publication of the study.
Access Criteria: Data access requests will be reviewed by external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Aryal UR, Vaidya A, Shakya-Vaidya S, Petzold M, Krettek A. Establishing a health demographic surveillance site in Bhaktapur district, Nepal: initial experiences and findings. BMC Res Notes. 2012 Sep 5;5:489. doi: 10.1186/1756-0500-5-489. PMID 22950751
- [Background] Nepal M, Pokharel B, Nepal P. Awareness and attitude regarding cardiovascular diseases among the adolescents studying in grade 12 in Makawanpur Multiple Campus in Nepal. Int J Heal Sci Res. 2021;11(5):261-8.
- [Background] Yadav K, Wagle R. Knowledge and attitude regarding major risk factors of cardiovascular diseases among 15-19 year old students of Kathmandu District. Heal Prospect. 2012;11:7-10.
- [Background] Aryal KK, Bista B, Khadka BB, Pandey AR, Mehta R, Jha BK, et al. Global School Based Student Health Survey Nepal-2015. Global School Based Student Health Survey Nepal. Nepal Health Research Council; 2015.
- [Background] Khanal MK, Mansur Ahmed MSA, Moniruzzaman M, Banik PC, Dhungana RR, Bhandari P, Devkota S, Shayami A. Prevalence and clustering of cardiovascular disease risk factors in rural Nepalese population aged 40-80 years. BMC Public Health. 2018 May 31;18(1):677. doi: 10.1186/s12889-018-5600-9. PMID 29855293
- [Background] Pearson TA, Palaniappan LP, Artinian NT, Carnethon MR, Criqui MH, Daniels SR, Fonarow GC, Fortmann SP, Franklin BA, Galloway JM, Goff DC Jr, Heath GW, Frank AT, Kris-Etherton PM, Labarthe DR, Murabito JM, Sacco RL, Sasson C, Turner MB; American Heart Association Council on Epidemiology and Prevention. American Heart Association Guide for Improving Cardiovascular Health at the Community Level, 2013 update: a scientific statement for public health practitioners, healthcare providers, and health policy makers. Circulation. 2013 Apr 23;127(16):1730-53. doi: 10.1161/CIR.0b013e31828f8a94. Epub 2013 Mar 21. No abstract available. PMID 23519758
- [Background] Eckel RH, Jakicic JM, Ard JD, de Jesus JM, Houston Miller N, Hubbard VS, Lee IM, Lichtenstein AH, Loria CM, Millen BE, Nonas CA, Sacks FM, Smith SC Jr, Svetkey LP, Wadden TA, Yanovski SZ, Kendall KA, Morgan LC, Trisolini MG, Velasco G, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 AHA/ACC guideline on lifestyle management to reduce cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S76-99. doi: 10.1161/01.cir.0000437740.48606.d1. Epub 2013 Nov 12. No abstract available. PMID 24222015
- [Background] Lichtenstein AH, Appel LJ, Vadiveloo M, Hu FB, Kris-Etherton PM, Rebholz CM, Sacks FM, Thorndike AN, Van Horn L, Wylie-Rosett J. 2021 Dietary Guidance to Improve Cardiovascular Health: A Scientific Statement From the American Heart Association. Circulation. 2021 Dec 7;144(23):e472-e487. doi: 10.1161/CIR.0000000000001031. Epub 2021 Nov 2. PMID 34724806